CLINICAL TRIAL: NCT01740609
Title: A Phase 1 Study To Evaluate The Safety, Tolerability, Immunogenicity, Pharmacokinetics And Pharmacodynamics Of Escalating Doses Of Pf-06342674 (RN168) In Healthy Volunteers
Brief Title: A Study To Assess The Safety Of PF-06342674 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B4351001
Record Dates: First submitted 2012-11-05; First posted 2012-12-04 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Phase 1; RN168; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2.0 (Experimental)
  Interventions: Biological: PF-06342674 Dose A; Biological: PF-06342674 Dose B; Biological: PF-06342674 Dose C; Biological: PF-06342674 Dose D; Biological: PF-06342674 Dose E; Biological: PF-06342674 Dose F; Biological: PF-06342674 Dose G; Biological: PF-06342674 Dose H; Biological: PF-06342674 Dose I; Biological: PF-06342674 Dose J

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1. Placebo
Biological: PF-06342674 Dose A — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose B — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose C — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose D — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose E — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose F — Single IV Dose
  Arms: 2.0
Biological: PF-06342674 Dose G — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose H — Single IV Dose
  Arms: 2.0
Biological: PF-06342674 Dose I — Single SC Dose
  Arms: 2.0
Biological: PF-06342674 Dose J — Single IV Dose
  Arms: 2.0

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of single escalating doses PF-06342674.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and female of non-childbearing potential subjects between the ages of 18 and 55.
* BMI between 18.5 to 32 kg/m2.
* Total body weight ≥40 kg and ≤120 kg.

Exclusion Criteria:

* Previous treatment with an antibody within 6 months prior to Day 1.
* Pregnant or nursing females; females of childbearing potential.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting or intolerable treatment related AEs | 60 days
Incidence of treatment emergent AEs | 60 days
Incidence of abnormal laboratory findings | 60 days
Changes from baseline in safety laboratory assessments | 60 days
Abnormal and clinically relevant changes in vital signs, blood pressure, and ECG parameters | 60 days
Incidence of anti-drug-antibodies | 60 days
Severity of treatment emergent AEs | 60 days
Causal relationship of treatment emergent AEs | 60 days

SECONDARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | 60 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 60 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 60 days
PK parameter estimates including T1/2. | 60 days
Systemic Clearance (CL) | 60 days
  CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Apparent Oral Clearance (CL/F) | 60 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 60 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4351001&StudyName=A%20Study%20To%20Assess%20The%20Safety%20Of%20PF-06342674%20In%20Healthy%20Volunteers